CLINICAL TRIAL: NCT04159935
Title: Investigating iLux Efficacy in Contact Lens Wearers With Evaporative Dry Eye Disease
Acronym: SHEEPDOG
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Cancelled due to COVID-19
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41401
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- iLux® treatment (Experimental): The treatment group will receive iLux® treatment at Visit 1 and will be reviewed 1- and 3-months after iLux® treatment.
  Interventions: Device: iLux® system
- Delayed iLux® treatment (Experimental): Delayed iLux® treatment provided after 1 month (i.e. 1 month of no treatment, administer treatment after 1 month). Review 1- and 3-months after iLux® treatment.
  Interventions: Device: iLux® system

INTERVENTIONS:
Device: iLux® system — Commercially available medical device intended for use by qualified eye care professionals to apply localized heat and pressure therapy to a patient's eyelids.

SUMMARY:
The purpose of this clinical trial is to investigate the efficacy of a single iLux® treatment in symptomatic CL wearers who have DED (according to the TFOS DEWS II diagnostic criteria), of the evaporative dry eye disease subtype (EDE).

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Is willing and able to follow instructions and maintain the appointment schedule;
4. Has been using the same CL type (brand, material and dimensions) for > 3 months;
5. Wears commercially available soft CLs on average >2 hours per day, 4-7 days per week;
6. Is willing to try to wear their habitual CLs on average ≥ 6 hours per day, 4-7 days per week and maintain this for the duration of their involvement in the study;
7. Demonstrates an acceptable lens fit of their habitual contact lenses;
8. Does not have contact lens discomfort due to contact lens fit, lens material or known solution compatibility issues, in the opinion of the investigator;
9. Has at least one month supply of their habitual contact lens products at the time of the screening visit;
10. Has a CLDEQ-8 score ≥ 12;
11. Has dry eye symptoms without CL wear (OSDI ≥ 13) and has at least one of the two following signs:

    1. Non-invasive tear break-up time (NITBUT) of < 10 seconds in at least one eye;
    2. Fluorescein staining: > 5 spots of corneal staining OR > 9 conjunctival spots OR lid wiper staining (≥ 2mm length, ≥ 25% width) in at least one eye;
12. Has a lipid layer thickness of ≤ 100 nm in both eyes;
13. A meibomian gland secretion score (MGS) of ≤ 15 for 15 glands of the lower lid in both eyes.

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has used any prescription systemic medications or topical treatments for MGD or dry eye for the past 30 days prior to the screening visit and not willing to stop using these for the study duration (excluding over-the-counter artificial tears, dietary supplements and ocular lubricants but includes warm compresses, eyelid massage, eyelid hygiene, manual meibomian gland expression, punctal plug insertion or punctal occlusion, intense pulsed light treatment of the face or eyelids);
3. Has previously received treatment with an eyelid thermal pulsation device;
4. Has a history of any of the following ocular (eye or eyelid) conditions or procedures in either eye within the past 90 days prior to the screening visit:

   1. Ocular trauma
   2. Chemical burns
   3. Ocular Herpes simplex or Herpes zoster infection
   4. Limbal stem cell deficiency
   5. Recurrent ocular inflammation (e.g. uveitis, iritis, scleritis, episcleritis, keratitis)
5. Has undergone ocular surgery (e.g. intraocular, oculoplastic, corneal or refractive surgery procedure) within the past 12 months prior to the screening visit;
6. Has permanent make-up or tattoos on their eyelids;
7. Has any other known active* ocular disease and/or infection in either eye including: cicatricial lid margin disease or severe (≥ grade 3) blepharitis; moderate to severe (grade 2-4) allergic, vernal or giant papillary conjunctivitis; a hordeolum or stye; ocular surface abnormality that may compromise corneal integrity (e.g. Grade 3 corneal fluorescein staining, recurrent corneal erosion, corneal epithelial defect, map dot fingerprint dystrophy, previously treated chemical burn);
8. Has an eyelid abnormality that affects normal lid function (e.g. entropion, ectropion, oedema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis);
9. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
10. Has any other condition that could compromise treatment or increase the risk of a procedure-related injury;
11. Is using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
12. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study;
13. Has a history of sensitivity to rapidly blinking lights or photosensitive epilepsy;
14. Is pregnant, lactating or planning a pregnancy (by verbal communication) at the time of enrolment;
15. Is aphakic;
16. Is a member of CORE directly involved in the study;
17. Has taken part in a clinical research study within the last 30 days. * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — Centre for Ocular Research & Education
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single site between November 2019 and March 2020. The first participant was enrolled on November 15, 2019 and the last participant was enrolled on March 4, 2020.
Pre-assignment Details: Of 28 enrolled participants, 8 met inclusion criteria and were randomized to treatment.
Period: Overall Study
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Started | 4 | 4
Month 1 Post-treatment | 3 | 3
Month 3 Post-treatment | 3 | 1
Completed | 3 | 1
Not Completed | 1 | 3
Not completed — Study terminated due to COVID-19 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | iLux® Treatment | Delayed iLux® Treatment | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.0 (19.6) | 30.3 (13.2) | 33.6 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 4 | 8
Standard Patient Evaluation of Eye Dryness Questionnaire score [Mean (Standard Deviation); unit: scores on a scale] — The Standard Patient Evaluation of Eye Dryness questionnaire is a dry eye questionnaire developed to assess the frequency (0-3 scale, with higher values indicating more frequent symptoms) and severity (0-4 scale, with higher values indicating more severe symptoms) of patient symptoms. The questionnaire reviews the presence of symptoms within the past 72 hours and past 3 months. Scores range from 0-28, with higher values indicating more severe dryness.
  scores on a scale | 14 (6.6) | 11.8 (3.8) | 12.9 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Standard Patient Evaluation of Eye Dryness (SPEED) Questionnaire Score From Baseline to 1 Month
Description: The mean change in dry eye symptoms from baseline based on the Standard Patient Evaluation of Eye Dryness (SPEED) questionnaire score was evaluated 1 month after iLux treatment. The SPEED questionnaire is a dry eye questionnaire developed to assess the frequency (0-3 scale, with higher values indicating more frequent symptoms) and severity (0-4 scale, with higher values indicating more severe symptoms) of patient symptoms. Scores range from 0-28. A higher SPEED score represents more frequent and/or more severe symptoms.
Time Frame: 1 month
Population: 1 participant in each arm lost to follow-up due to COVID-19.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 3 | 3
scores on a scale | 2.0 (1.7) | -2.0 (6.2)
Statistical Analysis 1: Comparison: iLux® Treatment vs Delayed iLux® Treatment; Test type: Other; p = 0.400, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Meibomian Gland Score at Baseline
Description: To determine the meibomian gland score, secretion characteristics of 15 meibomian glands along the lower eyelid were evaluated including five glands each in the temporal, central and nasal regions of the lower eyelid. For each gland, secretion characteristics were graded as 3 (clear liquid), 2 (cloudy liquid), 1 (inspissated/ toothpaste consistency) and 0 (no secretion). The total meibomian gland score is the sum of the grades for all 15 glands with a range between 0 and 45. A higher score reflects less meibomian gland dysfunction.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 4 | 4
scores on a scale | 10.5 (4.7) | 10.5 (4.1)
Statistical Analysis 1: Comparison: iLux® Treatment vs Delayed iLux® Treatment; Test type: Other; p = 0.057, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Meibomian Gland Score at 1 Month
Description: as for outcome 2
Time Frame: 1 Month
Population: 1 participant in each arm was lost to follow-up due to COVID-19.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 3 | 3
scores on a scale | 21.3 (11.7) | 20.3 (10.1)
Statistical Analysis 1: Comparison: iLux® Treatment vs Delayed iLux® Treatment; Test type: Other; p = 1.000, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Meibomian Gland Score at 3 Months
Description: as for outcome 2
Time Frame: 3 Months
Population: 2 participants in the iLux® treatment group were assessed remotely due to the COVID-19 shutdown. Meibomian gland score was unable to be assessed via a remote visit. 1 participant in the iLux® treatment group and 3 participants in the delayed iLux® treatment group were lost to follow-up due to COVID-19. Meibomian gland score was not assessed in the 1 person in the delayed iLux® treatment group that completed the study as per the protocol.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 1 | 0
score on a scale | 15 [15 to 15] |

5. Secondary Outcome: Comfortable Contact Lens Wear Time at Baseline
Description: Participants reported how long the contact lenses on average were comfortable (comfortable wear time).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 4 | 4
Hours per day | 4.3 (2.6) | 2.3 (1.0)
Statistical Analysis 1: Comparison: iLux® Treatment vs Delayed iLux® Treatment; Test type: Other; p = 0.400, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Comfortable Contact Lens Wear Time at 1 Month
Description: Participants reported how long the contact lenses on average were comfortable (comfortable wear time).
Time Frame: 1 Month
Population: 1 participant in each arm lost to follow-up due to COVID-19.
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 3 | 3
Hours per day | 7.0 (4.6) | 4.0 (2.0)
Statistical Analysis 1: Comparison: iLux® Treatment vs Delayed iLux® Treatment; Test type: Other; p = 0.400, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Comfortable Contact Lens Wear Time at 3 Months
Description: Participants reported how long the contact lenses on average were comfortable (comfortable wear time).
Time Frame: 3 Months
Population: Participants lost to follow-up due to COVID-19.
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 3 | 1
Hours per day | 9.0 (3.6) | 2
Statistical Analysis 1: Comparison: iLux® Treatment vs Delayed iLux® Treatment; Test type: Other; p = 0.500, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Pre-lens Tear Break-up Time at Baseline
Description: The pre-lens tear film is the layer of tears located on top of the contact lens (i.e., between the eye lid and the contact lens). The time required for a dry spot to appear on the contact lens surface after blinking is referred to as the pre-lens tear break-up time. Three measurements are taken and averaged together. A higher number represents a longer pre-lens tear break-up time.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 4 | 4
Seconds | 5.1 (2.9) | 4.0 (1.1)
Statistical Analysis 1: Comparison: iLux® Treatment vs Delayed iLux® Treatment; Test type: Other; p = 1.00, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Pre-lens Tear Break-up Time at 1 Month
Description: as for outcome 8
Time Frame: 1 Month
Population: 1 participant in each arm lost to follow-up due to COVID-19.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 3 | 3
Seconds | 5.8 (3.9) | 3.3 (1.3)
Statistical Analysis 1: Comparison: iLux® Treatment vs Delayed iLux® Treatment; Test type: Other; p = 0.400, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Pre-lens Tear Break-up Time at 3 Months
Description: as for outcome 8
Time Frame: 3 Months
Population: 2 participants in the iLux® treatment group had a remote visit due to the COVID-19 closure of the site. Pre-lens tear break-up time was unable to be assessed using a remote visit. 1 participant in the iLux® treatment group and 3 participants in the delayed iLux® treatment group were lost to follow-up due to COVID-19. Pre-lens tear break-up time was not assessed in the 1 person in the delayed iLux® treatment group that completed the study as per the protocol.
Measure: Mean (Full Range); unit: Seconds
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 1 | 0
Seconds | 5.6 [5.6 to 5.6] |

11. Secondary Outcome: Average Contact Lens Wear Time at Baseline
Description: Participants reported how long they wore their contact lenses on average per day (total wear time).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 4 | 4
Hours per day | 10.5 (3.7) | 7.3 (2.5)
Statistical Analysis 1: Comparison: iLux® Treatment vs Delayed iLux® Treatment; Test type: Other; p = 0.343, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Average Contact Lens Wear Time at 1 Month
Description: Participants reported how long they wore their contact lenses on average per day (total wear time).
Time Frame: 1 Month
Population: 1 participant in each arm lost to follow-up due to COVID-19.
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 3 | 3
Hours per day | 12.3 (5.5) | 8.0 (0.0)
Statistical Analysis 1: Comparison: iLux® Treatment vs Delayed iLux® Treatment; Test type: Other; p = 0.700, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Average Contact Lens Wear Time at 3 Months
Description: Participants reported how long they wore their contact lenses on average per day (total wear time).
Time Frame: 3 Months
Population: Participants lost to follow-up due to COVID-19.
Measure: Mean (Standard Deviation); unit: Hours per day
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
Number analyzed (Participants) | 3 | 1
Hours per day | 12.7 (4.2) | 8 (0)
Statistical Analysis 1: Comparison: iLux® Treatment vs Delayed iLux® Treatment; Test type: Other; p = 0.500, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: A maximum of 4 months
Description: Regular investigator assessment
Arm/Group | iLux® Treatment | Delayed iLux® Treatment
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

LIMITATIONS AND CAVEATS:
The study was cancelled due to COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT04159935/Prot_SAP_000.pdf